CLINICAL TRIAL: NCT06591052
Title: Acute Effects of Passive and Proprioceptive Neuromuscular Facilitation Stretching Techniques on Speed, Agility and Explosive Strength in Elite Youth Basketball Players: Randomized Controlled Study
Brief Title: Acute Effects of Passive and Proprioceptive Neuromuscular Facilitation Stretching Techniques in Youth Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ACetinkaya005
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Basketball Players; Stretching; Physical Performance
Keywords: Basketball players; passive stretching; PNF stretching
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Passive Group (Experimental): Passive stretching was administered to the hamstring, quadriceps, and calf muscles by the same physiotherapist for participants in the passive group.
  Interventions: Other: Passive stretching
- PNF group (Experimental): The "hold-relax" technique, a specialized method within PNF (Proprioceptive Neuromuscular Facilitation), was applied by the same physiotherapist to the hamstring, quadriceps, and calf muscles of the participants in the PNF group.
  Interventions: Other: PNF stretching

INTERVENTIONS:
Other: Passive stretching — The physiotherapist positioned each muscle in its maximum lengthened state and held it there for 30 seconds. This process was repeated three times, with a 30-second rest interval between each stretch of the different muscle groups.
  Arms: Passive Group
Other: PNF stretching — The physiotherapist initially positioned each muscle in its most extended state, similar to the positions used in passive stretching. In this extended position, the participants performed an isometric contraction against maximal resistance in the antagonist direction for 5-8 seconds. Following the isometric contraction, participants were instructed to actively relax, and after a 5-second waiting period to ensure complete relaxation, the movement range was passively increased. The new end point of the extended range of motion was held for 30 seconds. This stretching protocol was repeated three times for each muscle group, with a 30-second rest period between each stretch.
  Arms: PNF group

SUMMARY:
The aim of this clinical trial is to learn the acute effects of passive stretching and proprioceptive neuromuscular facilitation (PNF) stretching techniques on agility, speed and lower extremity explosive strength in young basketball players. It will also provide information about the comparison of two different stretching techniques. The main questions it aims to answer are:

Does passive stretching have positive acute effects on agility, speed and lower extremity explosive strength? Does PNF stretching have positive acute effects on agility, speed and lower extremity explosive strength? The acute effects of passive stretching and PNF stretching on agility, speed and lower extremity explosive strength will be compared.

Participants:

First tests were performed after the same warm-up program. Then, one of the two different stretching techniques was applied and the same tests were repeated immediately afterwards.

DETAILED DESCRIPTION:
The aim of this study was to examine the acute effects of static passive and proprioceptive neuromuscular facilitation (PNF) stretching techniques on agility, speed and lower extremity explosive power in youth basketball players. Twenty male basketball players were randomized as passive and PNF groups. A single session of technique was applied to each group. Outcome measurements consisted of the T Agility Test, 30-Meter Sprint Test, Standing Long Jump Test, and Lateral Jump Test.

ELIGIBILITY:
Inclusion Criteria:

* being male
* being between 14-18 years of age
* having at least 2 years of basketball experience
* participated in regular team training for at least 2 months
* having a body mass index of <29.9 kg/m2

Exclusion Criteria:

* presence of pain and/or history of injury in the lower extremity within the last 6 months
* history of orthopedic surgery of the lower extremity

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
T agility test | Immediately before and after the stretching intervention, assessed within a single session, approximately 30 minutes in total
  The T agility test is used to assess an athletes agility and ability to change direction quickly. The test is set up with four cones arranged in a T shape. The athlete starts at the base of the T and sprints forward to the second cone, then turns right and runs to the right cone, touching it. Next, they run to the left cone and touch it, return to the middle cone, and finally sprint back to the starting point. The time is recorded with a stopwatch, starting when the athlete begins and stopping when they return to the starting point. Lower times indicate better agility performance.

SECONDARY OUTCOMES:
30-meter sprint test | Immediately before and after the stretching intervention, assessed within a single session, approximately 30 minutes in total
  The 30-meter sprint test is used to measure an athletes speed over a short distance. The test is conducted on a flat, straight surface. The athlete starts in a standing position behind the starting line. On the command, they sprint as fast as possible for 30 meters. The time is recorded with a stopwatch, starting when the athlete begins their sprint and stopping when they cross the 30-meter line. Faster times indicate better sprinting speed.
Lateral long jump test | Immediately before and after the stretching intervention, assessed within a single session, approximately 30 minutes in total
  The lateral long jump test is used to measure an athletes explosive leg power. In the lateral jump test, the participant positioned the lateral edge of their dominant foot next to the starting line, assumed a squat position, and then executed a maximal jump to the side. The test was performed twice, and the distance between the medial side of the dominant foot and the starting line at the landing position was measured and recorded.
Standing long jump test | Immediately before and after the stretching intervention, assessed within a single session, approximately 30 minutes in total
  The standing long jump test is used to measure an athletes explosive leg power. The athlete stands behind a marked line with their feet shoulder-width apart. From a standing position, they bend their knees and swing their arms to jump forward as far as possible. The distance jumped is measured from the starting line to the nearest point of contact (usually the back of the heels) where the athlete lands. The best of three attempts is recorded. Longer jumps indicate greater lower body power.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Çetinkaya, Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No